CLINICAL TRIAL: NCT04939480
Title: Window of Opportunity Study of Preoperative Immunotherapy With Atezolizumab (Tecentriq®) in Local Head and Neck Squamous Cell Carcinoma (the PIONEER Trial)
Brief Title: Window of Opportunity Study of Preoperative Immunotherapy With Atezolizumab in Local SCCHN
Acronym: PIONEER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO39839
Record Dates: First submitted 2021-05-28; First posted 2021-06-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-08

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Pre-operative administration of atezolizumab 1200 mg followed by definitive resection of the tumor, followed by standard of care radiotherapy or radio-chemotherapy.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg intravenous solution

SUMMARY:
Targeting the PD-L1 pathway with atezolizumab has demonstrated objective responses across a broad range of malignancies including head and neck squamous cell carcinoma (SCCHN). MO39839 is a window of opportunity study investigating the feasibility, safety and postoperative complication rates of preoperative short time immunotherapy with atezolizumab in patients with local SCCHN. In the scope of MO39839 a comprehensive translational research program will be conducted to assess the potential effect of atezolizumab on dynamics in tumor immunity, and to identify and validate potential predictive and prognostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol. Written informed consent has to be obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations. If laboratory or imaging procedures were performed for alternate reasons prior to signing consent, these can be used for screening purposes with consent of the patient. However, all screening examinations and laboratory results must have been obtained within 14 days before first study drug administration (initial tumor imaging: within 28 days before first study drug administration).
2. Only patients for whom sufficient tumor material to be judged by the local investigator and which is of adequate quality can be included into the trial. Please refer to section 6.5 for further details on quantity and quality of tumor samples.
3. Histologically or cytologically proven SCCHN (cT1-4a, cN0-3, cM0) that is amenable to surgical resection with curative intent based on the decision of the local multidisciplinary tumor board.
4. Patients with relapse after primary radio(chemo)-therapy are allowed if a salvage surgery is possible (maximum 20%). Patients should have recovered from the effects of radiation: AE/sequelae should resolves to ≤ grade 2 (no minimum recovery period required).
5. Male or female, 18 years of age or older on day of signing informed consent
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
7. Life expectancy >12 weeks
8. Adequate hematologic and end-organ function, defined by laboratory test results, obtained within 14 days prior to initiation of study treatment
9. Women of childbearing potential: Should have a negative urine or serum pregnancy test within 14 days prior to receiving the first dose of study medication. Agreement to remain abstinent (refrain from heterosexual intercourse) or use a non-hormonal contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 5 months after last study drug administration

Exclusion Criteria:

1. Evidence of metastatic disease (M1)
2. cT4b Stage
3. Prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
4. Treatment with investigational therapy within 28 days prior to initiation of study treatment
5. Any anti-cancer therapy, including chemotherapy or hormonal therapy, within 4 weeks prior to initiation of study treatment
6. Bilateral pleural effusion
7. Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to Day 1, Cycle 1. Note: The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e. for adrenal insufficiency) and mineralocorticoids (e.g. fludrocortisone) is allowed
8. Treatment with a live-attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study, and for 5 months after the last dose of atezolizumab
9. Treatment with systemic immuno-stimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment
10. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation
11. Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
12. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
13. Uncontrolled tumor-related pain. Patients requiring narcotic pain medication must be on a stable regimen at study entry
14. Pregnant and lactating women
15. Acute toxicities from previous therapy that have not resolved to Grade ≤ 1, except for alopecia
16. Infections

    1. Positive human immunodeficiency virus (HIV): Known HIV+ patients may be included but must have:

       A stable regimen of highly active anti-retroviral therapy (HAART) No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests
    2. Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening followed by a negative HBV DNA test, are eligible for the study. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
    3. Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test at screening.

       The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
    4. Active tuberculosis
    5. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
    6. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
    7. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
17. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (see Appendix 12.1 for a more comprehensive list of autoimmune diseases and immune deficiencies) with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., no psoriatic arthritis) may be eligible provided that they meet the following conditions: Rash must cover less than 10% of the body surface area, disease is well controlled at baseline and only requires low potency topical steroids, and there are no acute exacerbations of underlying condition within the last 12 months (e.g. not requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency, or oral steroids)
18. Adverse events (AE) related to any previous radiotherapy, chemotherapy, targeted therapy or surgical procedure that have not resolved to Grade ≤1, except alopecia (any grade) and Grade 2 neuropathy
19. Prior allogeneic stem cell or solid organ transplantation
20. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computer tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
21. Active malignancy or a prior malignancy within the past 3 years. Patients with completely resected basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and patients with isolated elevation in prostate-specific antigen in the absence of radiographic evidence of metastatic prostate cancer are eligible for the study.
22. Any Grade 3 or higher hemorrhage or bleeding event within 28 days of Day 1 of Cycle 1
23. Increased corrected QT (QTc) interval (QTc > 470 ms)
24. Family history of long QT syndrome or other risk factors for torsades de pointes
25. History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to Day 1
26. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 6 months prior to Cycle 1 Day 1, severe cardiac arrhythmia requiring medication or severe conduction abnormalities, unstable arrhythmias, acute coronary syndromes (including unstable angina), or history of coronary angioplasty/stenting/bypass grafting within past 6 months.

    1. Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded
    2. patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
27. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
28. Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety
29. Participation in another clinical study within the last 3 months prior to inclusion or simultaneous participation in other clinical studies with an exception of studies evaluating radiological imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Effect of atezolizumab on tumor-infiltrating immune cells in resectable SCCHN | 4 weeks
  Percentage of patients with at least 2-fold increase of GzmB+/CD8+ T cells by immunohistochemistry (IHC) after 1 administration of atezolizumab between pre-treatment biopsy specimens and post-treatment resection specimens
Feasibility of preoperative short time immunotherapy | 3 weeks
  Number of patients with completion of pre-operative immunotherapy and resection of SCCHN

SECONDARY OUTCOMES:
Safety of preoperative short time immunotherapy | 58 days
  Number and grade of AEs (CTC AE v5.0)
Assessment of postoperative complication rates | 30 days
  Number and grade of AEs within 30 days postoperative (CTC AE v5.0)
To assess dynamics in tumor immunity | 21 days
  Changes (measured as the relative frequency within total tumor infiltrating leukocytes determined by CD45 marker) in tumor infiltrating CD66b, CD68, CD3, CD19, CD56 positive immune cells between day 1 (biopsy) and day 21 (surgery specimen). Frequency will be determined by immunofluorescence and software-based image analysis.
Characterization of changes in frequency of circulating immune cells | 58 days
  Changes (measured as the relative frequency within total circulating leukocytes determined by CD45 marker) in circulating CD66b, CD68, CD3, CD19, CD56 positive immune cells between day 1 and day 58. Frequency will be determined by flow cytometry.
Resectability after immunotherapy | 4 weeks
  Number of patients with R0 or R1 resection
Influence of immunotherapy on histo-morphological assessment | 21 days
  Changes of tumor-stroma ratio and total density of tumor infiltrating leukocytes between day 1 (biopsy) and day 21 (surgical specimen). Parameters will be assessed and quantified using immunofluorescence markers (EpCAM, cytokeratin, vimentin, CD45, DAPI) and digital pathology tools.
(optional) set up of a registry for follow up of patients and subsequent documentation of relapse free survival (RFS) rate and overall survival (OS) rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kasper-Virchow, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No